CLINICAL TRIAL: NCT03545386
Title: Randomized Trial of Fecal Microbiota Transplantation Versus Placebo for the Induction of Remission in Patients With Active Pouchitis
Brief Title: Fecal Microbiota Transplantation for Pouchitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4702
Record Dates: First submitted 2018-05-10; First posted 2018-06-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT (Experimental)
  Interventions: Other: Fecal microbiota transplantation
- Placebo (Placebo Comparator)
  Interventions: Other: Placebos

INTERVENTIONS:
Other: Fecal microbiota transplantation — Stool from healthy donor administered via enema
  Arms: FMT
Other: Placebos — Saline with food coloring administered via enema
  Arms: Placebo

SUMMARY:
This is a randomized double-blind placebo controlled trial involving a single centre (McMaster University) recruiting patients from Hamilton, ON and the surrounding regions, to evaluate whether fecal microbiota transplantation once weekly for six weeks increases the remission rate compared to placebo in patients with active pouchitis.

DETAILED DESCRIPTION:
Patients with ulcerative colitis (UC) may undergo colectomy due to a variety of reasons, including medically refractory disease or dysplastic changes of the colon. Ileal-pouch anal anastomosis is often offered to these patients. Unfortunately the pouch commonly develops inflammation, known as pouchitis, which is the most common complication of this procedure and occurs in approximately 50% of patients, with the majority of these patients having multiple episodes.

Although the exact cause of pouchitis is not clear, it is felt that fecal bacteria may be implicated in the cause. Studies have demonstrated changes in the fecal contents of patients with pelvic pouches compared to those with end ileostomies, with higher concentrations of Bacteroides and stool anaerobes identified in those patients with pelvic pouches. Antibiotics are a mainstay of treatment for pouchitis, with randomized controlled trials demonstrating response rates of 70-85% to metronidazole or ciprofloxacin for treatment of acute pouchitis. Unfortunately, recurrent use of systemic antibiotics is associated with adverse events and development of antibiotic resistance.

Fecal Microbiota Transplantation (FMT) is the administration of the supernatant component of stool and water mixture from a healthy screened donor. The donors are screened for numerous infections and pathogens prior to being accepted as donors. FMT has been advocated for some colonic disorders; however it is primarily used in recurrent/refractory Clostridium difficile infections (CDI). A case series from McMaster of over 100 patients and have shown that approximately 90% of patients with recurrent CDI have been cured with FMT. The rationale is that the aberrant colonic microbiome can be replaced with a normal healthy microbiome from a donor. A similar rationale has been applied to ulcerative colitis, and a recent systematic review and meta-analysis conducted by the investigators demonstrated FMT is associated with improved clinical remission and endoscopic healing compared to placebo. It seems possible that changing the intestinal flora in patients with pouchitis could also return the mucosa to a healthy state.

The investigators have conducted the world's first randomized trial of fecal transplant therapy to determine its efficacy and safety in patients with active UC. The investigators found that fecal transplants given once per week for 6 weeks resolved the inflammation in 24% of patients with active UC compared to 5% with placebo. There has been no randomized control trial evaluating the efficacy of FMT for treatment of pouchitis. An initial case series of 8 patients did not find treatment with one administration of FMT via nasogastric administration to be associated with any improvement in clinical response. However a subsequent case series found improvement in 4 out of 5 patients with chronic pouchitis who had multiple FMT treatments over 3-4 weeks. The investigators will conduct a randomized trial at a single centre (McMaster University) comparing fecal transplant therapy (from a healthy donor) versus placebo for six weeks for induction of remission in patients with active pouchitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or over
2. Active pouchitis defined as PDAI of 7-18 points
3. Females of child bearing potential must be willing and able to use acceptable contraception as per Appendix III. II. b. Toxicity section of the Health Canada Guidance

Exclusion Criteria:

1. Participating in another clinical trial
2. Unable to give informed consent
3. Severe comorbid medical illness
4. Concomitant Clostridium difficile infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Remission of pouchitis, defined as a pouchitis disease activity index (PDAI) score of <7, with a decreased from baseline PDAI score of 3 points | 7 weeks
  Comparison between FMT and placebo arms in remission rates

SECONDARY OUTCOMES:
compliance of patients who receive FMT | 7 weeks
  Measurement of retention rate of patients who receive FMT
compare the fecal microbiome in pouchitis patients in remission versus still active at the end of the trial. | 7 weeks
  Analysis of changes using 16S rRNA to look at changes in the bacterial profiles of patients who respond to FMT compared to those who do not

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No